CLINICAL TRIAL: NCT06696001
Title: Interbrain Synchronization of the Therapist-Client Dyad in Psychotherapy: Pilot EEG Study in Students With Mild-Moderate Depression Symptoms
Brief Title: Neuroscience of Psychotherapy for Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Foundation of Hope, North Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-1422
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Depression
Keywords: EEG; Hyperscanning; Therapeutic Alliance; Psychoeducation; behavioral activation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: There are two interventions that the participants will randomly be assigned to. Each participant will only complete one of these two interventions during their duration in the study.
Who Masked: Participant
Masking Description: The research assistants and personnel will be aware of the randomized intervention for each participant since this will be stored on an encrypted spreadsheet with a password. The participants will be made aware that they will be randomized to a group, however, they will not know what intervention they have been assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducation (Active Comparator): Psychoeducation will be used in this study as a control condition. The 60 minute session will be structured to provide general educational information on depression and evidence-based strategies to reduce symptoms. The information will be presented in generic format and will not be tailored to be client-specific.
  Interventions: Behavioral: Psychoeducation
- Behavioral Activation (Experimental): Behavioral Activation (BA) is a psychotherapy modality that can be used to treat depression. The 60 minute session of BA is designed to actively engage with the client in creating personalized goals and ways in which maladaptive coping mechanisms maintaining depression can be addressed and replaced with increased exposure to positive reinforcement.
  Interventions: Behavioral: Behavioral Activation

INTERVENTIONS:
Behavioral: Psychoeducation — For the psychoeducation session, the focus is for the therapist to engage with the client regarding mental health broadly without a targeted effort to reinforce therapeutic alliance or to offer individualized guidance or techniques. The session will provide educational information on depression, depression symptoms and known causes, and strategies to reduce depression symptoms. The content will be delivered in a fashion to avoid individualization and psychotherapeutic exchange. The elements will focus on components of Cognitive Behavioral Therapy (CBT), differentiating between thoughts and feelings, common cognitive shortcuts, and the connection between behavior and emotion.
  Arms: Psychoeducation
Behavioral: Behavioral Activation — Behavioral Activation (BA) is a psychotherapy treatment modality used for depression and focuses on replacing maladaptive coping mechanism that reinforce depressive symptoms with adaptive coping mechanisms to increase exposure to positive reinforcement. The treatment will consist of the following elements: Introduction to establish concept of positive reinforcement and build rapport, identification of client-centered values, individualized values-based activity planning and scheduling, and developing adaptive coping strategies for the future.
  Arms: Behavioral Activation

SUMMARY:
The goal of this study is to learn the extent to which client-therapist brain activity may synchronize during a psychosocial intervention for depression symptoms.

The study will compare behavioral activation, a client-centered type of cognitive-behavioral therapy, to psychoeducation which delivers information on strategies to recover from depression symptoms.

Participants will answer questions about their mental and physical health, attend one psychosocial intervention session receiving either Behavioral Activation or Psychoeducation with simultaneous brain activity measurement and complete follow up surveys two weeks and one month following the intervention.

DETAILED DESCRIPTION:
This is a pilot study to investigate the neuroscience of a single-session psychosocial intervention for depression symptoms. Brain activity is measured with EEG in both research participant and therapist. Participants will fill in questionnaires about their depression symptoms and experience during the psychosocial intervention.

ELIGIBILITY:
Inclusion Criteria for participants/clients:

* Between ages 18 and 30
* Full-time student status (undergraduate, graduate, and professional)
* Experience mild to moderate depressive symptoms as determined by the Beck Depression Inventory (score: 14-28)
* Capacity to understand study procedures (informed consent)
* Ability to speak and understand English
* Willingness to comply with study procedures

Inclusion Criteria for therapists:

* Ages 18 or older
* Qualification to administer therapy (decided by the Principal Investigator)
* Capacity to understand the study procedures (informed consent)
* Speak and understand English
* Willingness to comply with study procedures

Exclusion Criteria for participants/clients:

* Active, Current Suicidal ideation as determined by the Columbia-Suicide Severity Rating Scale (C-SSRS) in the past month
* Past suicidal attempt (lifetime)
* Recently initiated psychotherapy (past month)
* Elevated psychosis risk based on self-report prodromal questionnaire - brief version (PQ-B) or self-reported diagnosis of psychotic disorder by mental health provider
* Positive screen for autism spectrum disorder based on the self-report autism quotient (AQ-10) or self-reported diagnosis of autism spectrum disorder by mental health provider,
* Daily intake of benzodiazepine of >20 mg diazepam milligram equivalent
* Inability to give informed, voluntary, written consent to participate
* Inability to effectively communicate in English as determined by interaction with study personnel
* Anything else that in the assessment of the study team is not conducive to the successful completion of the study requirements.

There are no exclusion criteria for therapists

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Inter-brain phase synchronization in Alpha frequency band via Phase Locking Value | During the interventional session, approximately 60 minutes
  Inter-brain synchronization will be calculated for the Alpha frequency band via phase locking value during the interventional session for both study arms and will be used to assess any potential differences in Alpha frequency inter-brain synchronization between groups
Inter-brain phase synchronization in Theta frequency band via Phase Locking Value | During the interventional session, approximately 60 minutes
  Inter-brain synchronization will be calculated for the theta frequency band via phase locking value during the interventional session for both study arms and will be used to assess any potential differences in Theta frequency inter-brain synchronization between groups

SECONDARY OUTCOMES:
Directed inter-brain connectivity in theta frequency band via Granger Causality | During the intervention session, approximately 60 minutes
  The Granger causality test is a statistical hypothesis test that helps decide whether one time series can predict another and will be used to determine directed inter-brain connectivity. Granger causality will be calculated in the Theta frequency band during the interventional session for the Behavioral Activation arm to compare the direction of the connectivity as a function of the therapeutic elements.
Directed inter-brain connectivity in the Alpha frequency band via Granger Causality | During the intervention session, approximately 60 minutes
  The Granger causality test is a statistical hypothesis test that helps decide whether one time series can predict another and will be used to determine directed inter-brain connectivity. Granger causality will be calculated in the Alpha frequency band during the interventional session for the Behavioral Activation arm to compare the direction of the connectivity as a function of the therapeutic elements.
Correlation between Inter-brain Phase Synchronization in Alpha frequency band via phase locking value and change in depression symptoms via Beck Depression Inventory II (BDI) total score | Baseline Up to 4 weeks post-intervention session
  Alpha frequency band phase locking values calculated at the interventional session will be correlated with difference scores on Beck's Depression Inventory II from baseline to 4 weeks post intervention. The Beck's Depression Inventory is a 21-item instrument that measures characteristics and symptoms of depression. Possible scores range from 0-63, with lower scores indicating a better outcome with decreased symptoms of depression. Total difference scores on the BDI will be correlated with inter-brain phase synchronization to determine if there is a significant relationship between inter-brain phase synchronization in the alpha frequency band and change in depression symptoms 4 weeks post-intervention from baseline.
Correlation between Inter-brain Phase Synchronization in Theta frequency band via phase locking value and change in depression symptoms via Beck Depression Inventory II total score | Baseline Up to 4 weeks post-intervention session
  Theta frequency band phase locking values calculated at the interventional session will be correlated with difference scores on Beck's Depression Inventory II from baseline to 4 weeks post intervention. The Beck's Depression Inventory is a 21-item instrument that measures characteristics and symptoms of depression. Possible scores range from 0-63, with lower scores indicating a better outcome with decreased symptoms of depression. Total difference scores on the BDI will be correlated with inter-brain phase synchronization to determine if there is a significant relationship between inter-brain phase synchronization in the alpha frequency band and change in depression symptoms 4 weeks post-intervention from baseline.

OTHER OUTCOMES:
Correlation between inter-brain phase synchronization in theta frequency band via Phase Locking Value and therapeutic alliance via score on the Working Alliance Inventory (WAI) | immediately post-intervention
  The correlation between inter-brain phase synchronization in the theta frequency band and therapeutic alliance will be calculated using Pearson's Correlation Coefficient. Pooled Phase Locking value for each study arm will be correlated with pooled scores on the Working Alliance Inventory Short Form-Revised, a 12 item measure with a minimum score of 12 and a maximum score of 60. Both measures being correlated are collected at the immediately post-intervention.
Correlation between inter-brain phase synchronization in alpha frequency band via Phase Locking Value and therapeutic alliance via score on the Working Alliance Inventory (WAI) | immediately post-intervention
  The correlation between inter-brain phase synchronization in the alpha frequency band and therapeutic alliance will be calculated using Pearson's Correlation Coefficient. Pooled Phase Locking value for each study arm will be correlated with pooled scores on the Working Alliance Inventory Short Form-Revised, a 12 item measure with a minimum score of 12 and a maximum score of 60. Both measures being correlated are collected at the immediately post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, Principal Investigator — Carolina Center for Neurostimulation
Locations (1):
- Carolina Center for Neurostimulation, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: Beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, REB and an executed a data use/sharing agreement with UNC.

REFERENCES:
- [Background] Kazdin AE. Understanding how and why psychotherapy leads to change. Psychother Res. 2009 Jul;19(4-5):418-28. doi: 10.1080/10503300802448899. PMID 19034715
- [Background] Wampold BE. How important are the common factors in psychotherapy? An update. World Psychiatry. 2015 Oct;14(3):270-7. doi: 10.1002/wps.20238. PMID 26407772
- [Background] Hougaard E. The therapeutic alliance--a conceptual analysis. Scand J Psychol. 1994 Mar;35(1):67-85. doi: 10.1111/j.1467-9450.1994.tb00934.x. PMID 8191262
- [Background] Safran JD, Muran JC. Resolving therapeutic alliance ruptures: diversity and integration. J Clin Psychol. 2000 Feb;56(2):233-43. doi: 10.1002/(sici)1097-4679(200002)56:23.0.co;2-3. PMID 10718606
- [Background] Dumas G, Nadel J, Soussignan R, Martinerie J, Garnero L. Inter-brain synchronization during social interaction. PLoS One. 2010 Aug 17;5(8):e12166. doi: 10.1371/journal.pone.0012166. PMID 20808907